CLINICAL TRIAL: NCT03983460
Title: Dupilumab Impact on Skin Resident Memory T Cells
Acronym: DupiTrem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association pour la Recherche Clinique et Immunologique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18082A0002
Record Dates: First submitted 2019-05-21; First posted 2019-06-12 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Betamethasone Valerate; Biopsy; Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dupimulab arm (Experimental): At Day 0, patients will receive Dupilumab treatment. The recommended dose of Dupilumab for adult patients is an initial dose of 600mg followed by 300mg given every two weeks administered as subcutaneous injection. Dupilumab could be self-administered by subcutaneous injection into thigh or abdomen or injected in the upper arm in case of administration by the patient's caregiver. It is recommended to rotate the injection site with each injection.
  At the end of treatment period, patient with AD IGA >1 will stop the study and patient with AD IGA≤1 will enter in a 3 months-follow-up period. During this period, they will stop treatment initiated at Day 0 and apply rescue TCS if appearance of AD lesion within 3 months. Patients will note in their diary the applications of rescue TCS. The relapse is defined as the necessity to apply TCS rescues.
  Interventions: Drug: Dupilumab; Procedure: Biopsies; Procedure: Skin prick-test; Procedure: Blood sample collection
- Optimized TCS treatment arm (Active Comparator): At Day 0, patients will receive topical corticosteroid treatment (TCS) adapted to the AD severity (potent and very potent TCS) with a personal therapeutic education for treatment optimization. It will be asked to perform, every day, an application of topical corticosteroid (TCS) (betamethasone valerate cream 0.1%, and if not active, clobetasol propionate cream 0.05%) on active lesions. Once the AD lesion is cleared, the patients will continue to apply TCS on healed lesions, twice a week until the end of the treatment period to prevent relapse.
  At the end of treatment period, patient with AD IGA >1 will stop the study and patient with AD IGA≤1 will enter in a 3 months-follow-up period. During this period, they will stop treatment initiated at Day 0 and apply rescue TCS if appearance of AD lesion within 3 months. Patients will note in their diary the applications of rescue TCS. The relapse is defined as the necessity to apply TCS rescues.
  Interventions: Drug: Optimized TCS treatment; Procedure: Biopsies; Procedure: Skin prick-test; Procedure: Blood sample collection

INTERVENTIONS:
Drug: Dupilumab — Each single used prefilled syringe contains 300 mg of Dupilumab in 2 mL solution (150mg/mL) Dupilumab is a fully human monoclonal antibody against interleukin (IL)-4 receptor alpha that inhibits IL-4/IL-13 signaling, produced in Chinese Hamster Ovary (CHO) cells by recombinant DNA technology.
  Arms: Dupimulab arm
Drug: Optimized TCS treatment — Application of betamethasone valerate 0.1% (Betneval 0.1% cream), a potent topical corticosteroid, and if not active, application of clobetasol propionate 0.05% (Dermoval 0.05% cream), a very potent topical corticosteroid. TCS treatment will be associated with a personal therapeutic education for treatment optimization.
  Other Names: Betamethasone valerate 0.1% and Clobetasol propionate 0.05%
  Arms: Optimized TCS treatment arm
Procedure: Biopsies — Four skin biopsies (5 mm diameter) and ten microbiopsies (2 & 3 mm diameter) will be performed according the following schedule:
  * Day 0
    * a 5 mm section biopsy from a non-lesional skin
    * a 5 mm section biopsy from an active lesion
    * a 3 mm section microbiopsies from a non-lesional skin
    * a 3 mm section microbiopsies from an active lesion
    * a 2 mm section microbiopsies from a non-lesional skin
    * a 2 mm section microbiopsies from an active lesion
  * Day 28
    * a 5 mm section biopsy on improved/healed lesion
    * a 3 mm section microbiopsies on improved/healed lesion
    * a 2 mm section microbiopsies from non lesional skin identified at V1
    * a 2 mm section microbiopsies on improved/healed lesion
  * Day 168
    * a 5 mm section biopsy on improved/healed lesion
    * a 3 mm section microbiopsies on improved/healed lesion
    * a 2 mm section microbiopsies from non-lesional skin identified at V1
    * a 2 mm section microbiopsies on improved/healed lesion
Procedure: Skin prick-test — Skin prick test is a method for medical diagnosis of allergy consisting in introducing a small amount of an allergen into the patient's skin. The allergen penetrates the epidermis by pricking the skin with a pin.
  Skin Prick test for Derp and Derf will be performed at Day 0, preferentially on the forearms, avoiding lesional areas.
  For the results interpretation, the two allergen Derp/Derf will be compared to 2 controls:
  * Negative control : saline solution
  * Positive control : histamine solution
  Positive criteria of prick tests results are:
  * Positive control's diameter ≥ 3mm
  * And negative control's diameter < 3 mm
  * And tested allergen with wheal ≥ positive control, i.e. 3mm
Procedure: Blood sample collection — A 50ml blood sample will be collected by venipuncture at Day 0, Day 28 and Day 168.
  More specifically a 40 ml blood sample will be drawn on heparinized tubes for immunophenotyping and a 10 mL on serum blood collection tube for analysis of AD biomarkers by mass cytometry and ELISA.

SUMMARY:
The main objective of the study consists in characterizing the immune cells that are present/persist in the skin and the blood of atopic dermatitis (AD) patients treated with Dupilumab, as well as with potent/very potent topical corticosteroids (TCS: betamethasone valerate cream 0.1% or clobetasol propionate cream 0.05%). A specific attention will be paid on the presence/persistence of skin Trm and ILCs.

The study population will consist of 20 adult patients suffering from moderate to severe Atopic Dermatitis and eligible for Dupilumab treatment. (Patients should have inadequate response, intolerance or contraindication to systemic anti-inflammatory treatments).

This is an exploratory, prospective, single-site, randomized, open labeled study. There is a treatment period of 168 days (24 weeks) and a post-treatment follow-up period of maximum 102 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject over 18 years of age
* Subject able to read, understand and give documented informed consent
* Subject willing and able to comply with the protocol requirements for the duration of the study
* Subject with health insurance coverage according to local regulations
* For woman with childbearing potential :

  * Use of a highly effective method of birth control from at least 1 month prior to study enrollment until the last visit
  * Negative urine pregnancy test at inclusion visit A highly effective method of birth controlled is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, combined oral contraceptives, intrauterine device, double barrier methods (e.g. condom with spermicide), sexual abstinence or vasectomized partner. Woman with no childbearing potential is defined as: woman with amenorrhea for at least 12 months (without an alternative medical cause); woman who had undergone a permanent sterilization method (eg bilateral tubal occlusion which includes tubal ligation procedures, hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy.
* Subject diagnosed with moderate-to-severe AD, defined as SCORAD≥20 and/or EASI≥7 (Eichenfield et al., 2014)
* Subject with AD involvement of 10% (or more) Body Surface Area (BSA) according to component A of SCORAD
* Subject with I, II, III or IV skin phototype (according to Fitzpatrick scale)
* Subject accepting skin prick-tests and skin biopsies
* Subject having a least one non lesional area on the body (off head and neck, feet and hands)
* Subject eligible for systemic treatment
* Failure, intolerance or contraindication to available systemic treatments (i.e. cyclosporine/methotrexate)

Exclusion Criteria:

* Pregnancy or breast-feeding women, or planning to become pregnant or breastfeed during the study
* Women unwilling to use adequate birth control, if of reproductive potential and sexually active.
* Subject currently experiencing or having a history of other concomitant skin conditions that would interfere with evaluation of AD
* History of allergic reaction to local anesthetic product
* History of wound healing disorders (e.g. hypertrophic scars, keloids)
* Subject with known active infection to HBV, HCV or HIV
* Subject with known helminth infection
* Subject with known blood dyscrasia
* Subject having an allergen immunotherapy within 3 months before study
* Subject treated by antihistamine 5 days before study. Please note, antihistamine administered to treat allergic rhino conjunctivitis is allowed after V1.
* Subject treated with an investigational drug within 8 weeks or within 5 half-life (if known), whichever is longer, before the baseline visit
* Subject treated with cyclosporine, methotrexate oral corticosteroids, azathioprine, mycophenolate mofetil, and/or any other systemic immunosuppressor/immunomodulator within 4 weeks before the study
* Subject treated by a biologic therapy within 5 half-life before the study
* Subject treated with ultraviolet therapy within 4 weeks before study
* Subject treated with a live (attenuated) vaccine within 12 weeks before baseline visit
* Subject having a planned surgery during the study
* Subject presenting clinically significant medical disease that is uncontrolled despite treatment that is likely, in the opinion of the investigator, to impact patient's ability to participate in the study or to impact the study efficacy or safety assessments
* Subject with any additional condition that, in the opinion of the investigator, may interfere with the assessment or put the subject at risk
* Linguistic or mentally incapacity to sign the consent form
* Subject protect by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated)
* Subject in an exclusion period from a previous study or who is participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
To assess the change of the number (per biopsy or per mL of blood) and/or frequency (among live hematopoietic cells CD45+) of immune cells that are present in the skin and the blood of AD patients after Dupilumab or TCS treatment. | At Day 0, Day 28 and Day 168.
  In this exploratory study, comprehensive immunophenotyping investigations will be conducted on the immune cells extracted from blood, and from the lesional, healed and non lesional skin biopsies of each patient. Capitalizing on the use of mass cytometry technology, which allows comprehensive analysis of 35-40 different markers on the same cell, we will establish a precise mapping of immune cells that circulate or infiltrate/persist the different lesions.
  A specific focus will determine the frequency/number of Trms and ILCs inside the skin, notably type-2 Trms (such as IL-4/IL-13 producing TH2) and ILC2.

SECONDARY OUTCOMES:
To investigate correlations between each immunological parameter and each clinical score as a continuous quantitative variable, as well as each immunological parameter and quality of life index as a continuous quantitative variable. | At Day 0, Day 28 and Day 168
  In order to determine the immunological parameters associated with the clinical state of patients (measured using IGA, EASI, SCORAD, lesional area score and life quality index), the following procedure will be done for each clinical score, and at each time. First, the correlation between the clinical score and each immunological parameter will be tested using linear regression models, including the type of treatment as a co-variable (one model for each immunological parameter). Then, a multiple linear regression model will be performed, where explanatory variables will include the treatment as well as some of the immunological parameters, based on statistical considerations as well as on clinical considerations. Immunological parameters with p-value<0.05 from the multiple linear regression model will be considered as significantly associated with the clinical state of patients.
To investigate correlations between each immunological parameter and change in clinical score as a qualitative variable with 2 modalities as well as each immunological parameter and quality of life index, as a qualitative variable with 2 modalities. | At Day 28 and Day 168.
  In order to determine the immunological parameters associated with the clinical efficacy of Dupilumab and TCS treatments (measured using IGA, EASI, SCORAD and life quality index considered as qualitative variables with two modalities: good or bad responders), the following procedure will be done for each clinical score, and at each time. First, the correlation between the clinical score and each immunological parameter will be tested using logistic regression models, including the type of treatment as a co-variable (one model for each immunological parameter). Then, a multiple logistic regression model will be performed, where explanatory variables will include the treatment as well as some of the immunological parameters, based on statistical considerations as well as on clinical considerations. Immunological parameters with p-value<0.05 from the multiple logistic regression model will be considered as significantly associated with the clinical state of patients.
To investigate correlations between each immunological parameter and the development of new AD lesions in the 3 following months, as well as each immunological parameter and the interval of time between the end of treatment and AD relapse. | At Day 0, Day 28,Day 168 and during the 3 months follow-up period.
  In order to determine the immunological parameters associated with the development of new AD lesions, a logistic regression model, will be used for each immunological parameter and at each time. Then, a multiple logistic regression model will be performed for each time. Immunological parameters with p-value<0.05 from the multiple regression model will be considered as significantly associated with the clinical state of patients. In order to determine the correlation between the immunological parameters and the interval of time between the end of treatment and AD relapse, a linear regression model, will be used for each immunological parameter and at each time. Then, a multiple regression model will be performed for each time. Immunological parameters with p-value<0.05 from the multiple regression model will be considered as significantly associated with the clinical state of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Allergologie et Immunologie Clinique - Hôpital Lyon Sud, Pierre-Bénite, France